CLINICAL TRIAL: NCT06859554
Title: Assessing the Therapeutic Efficacy and Safety Profile of Glyceryl Trinitrate (GTN) and Nifedipine Ointments in Acute Anal Fissure Treatment: A Parallel-arm Clinical Trial
Brief Title: Efficacy and Safety of GTN vs. Nifedipine in Acute Anal Fissure: A Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hafiz Muhammad Hamza (Other)
Collaborators: Federal Government Polyclinic (Postgraduate Medical Institute) (Other)
Responsible Party: Sponsor-Investigator, Hafiz Muhammad Hamza, House Officer, Foundation University School of Health Sciences, Federal Government Polyclinic (Postgraduate Medical Institute)
Organization: Federal Government Polyclinic (Postgraduate Medical Institute) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FGPC.1/12/2024
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-02

CONDITIONS: Acute Anal Fissure; Anal Pain; Anorectal Disorders; Sphincter Spasm
Keywords: Anal fissure treatment; Glyceryl Trinitrate (GTN); Nifedipine ointment; Randomized controlled trial (RCT); Pain relief in anal fissures
MeSH Terms: conditions — Rectal Diseases | interventions — Nitroglycerin; Ointments; Nifedipine

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, parallel-arm clinical trial evaluating the efficacy and safety of GTN (0.2% and 0.4%) versus Nifedipine (0.2% and 0.5%) in the treatment of acute anal fissures.
Who Masked: Participant, Investigator
Masking Description: Participants do not know which specific treatment they are receiving, and investigators assessing outcomes are also blinded. However, care providers and data analysts are aware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: GTN 0.2% (Active Comparator): Participants in this arm will apply 0.2% Glyceryl Trinitrate (GTN) ointment twice daily for four weeks. The primary goal is to assess its efficacy in healing acute anal fissures and symptom relief while monitoring for side effects such as headaches and dizziness.
  Interventions: Drug: Glyceryl Trinitrate (GTN) 0.2% Ointment
- Arm 2: GTN 0.4% (Active Comparator): Participants in this arm will apply 0.4% Glyceryl Trinitrate (GTN) ointment twice daily for four weeks. This higher concentration aims to determine the dose-dependent efficacy and side effect profile compared to 0.2% GTN
  Interventions: Drug: Glyceryl Trinitrate (GTN) 0.4% Ointment
- Arm 3: Nifedipine 0.2% (Active Comparator): Participants in this arm will apply 0.2% Nifedipine ointment twice daily for four weeks. The study will evaluate its effectiveness in fissure healing, pain relief, and incidence of adverse effects such as local irritation or hypotension.
  Interventions: Drug: Nifedipine 0.2% Ointment
- Arm 4: Nifedipine 0.5% (Active Comparator): Participants in this arm will apply 0.5% Nifedipine ointment twice daily for four weeks. This higher concentration will assess whether increased potency provides superior symptom resolution and healing rates while monitoring potential side effects.
  Interventions: Drug: Nifedipine 0.5% Ointment

INTERVENTIONS:
Drug: Glyceryl Trinitrate (GTN) 0.2% Ointment — Participants will apply 0.2% Glyceryl Trinitrate (GTN) ointment to the anal region twice daily for four weeks. GTN functions as a nitric oxide donor, reducing internal anal sphincter tone to improve blood flow and promote fissure healing. The study aims to assess its effectiveness in symptom relief, fissure healing, and associated side effects such as headaches and dizziness.
  Other Names: GTN 0.2%; Nitroglycerin 0.2% Ointment
  Arms: Arm 1: GTN 0.2%
Drug: Glyceryl Trinitrate (GTN) 0.4% Ointment — Participants will apply 0.4% Glyceryl Trinitrate (GTN) ointment twice daily for four weeks. This increased concentration aims to determine dose-dependent efficacy and adverse effects in treating acute anal fissures. GTN acts by relaxing smooth muscle, decreasing sphincter tone, and enhancing mucosal blood flow to promote healing.
  Other Names: GTN 0.4%; Nitroglycerin 0.4% Ointment
  Arms: Arm 2: GTN 0.4%
Drug: Nifedipine 0.2% Ointment — Participants will apply 0.2% Nifedipine ointment twice daily for four weeks. Nifedipine, a calcium channel blocker, reduces sphincter tone by inhibiting calcium influx into smooth muscle cells, leading to improved fissure healing. This arm will assess its effectiveness in symptom relief and healing rates, with a focus on side effects such as local irritation or hypotension.
  Other Names: Nifedipine Gel 0.2%; Nifedipine 0.2%
  Arms: Arm 3: Nifedipine 0.2%
Drug: Nifedipine 0.5% Ointment — Participants will apply 0.5% Nifedipine ointment twice daily for four weeks. This higher concentration is used to evaluate whether increased potency provides superior symptom resolution and healing rates compared to 0.2% Nifedipine. The study will also assess any potential adverse effects, including local irritation, dizziness, and hypotension.
  Other Names: Nifedipine Gel 0.5%; Nifedipine 0.5%
  Arms: Arm 4: Nifedipine 0.5%

SUMMARY:
The goal of this clinical trial is to compare the therapeutic efficacy and safety profile of Glyceryl Trinitrate (GTN) and Nifedipine ointments in the treatment of acute anal fissures in adults. The main questions it aims to answer are:

Which ointment is more effective in promoting fissure healing and symptom relief? What are the adverse effects associated with each treatment? Researchers will compare GTN and Nifedipine ointments to determine which provides better symptom resolution with fewer side effects.

Participants will:

Apply GTN or Nifedipine ointment topically twice daily for four weeks Attend follow-up visits for symptom assessment and adverse effect monitoring

DETAILED DESCRIPTION:
Background and Rationale:

Anal fissures are painful linear tears in the anoderm, commonly caused by trauma from hard stool passage, leading to increased internal anal sphincter tone and ischemia. Acute fissures typically heal within six to eight weeks, while chronic fissures persist beyond this period. First-line treatment includes non-surgical options such as topical pharmacotherapy to reduce sphincter spasm and improve mucosal blood flow.

Glyceryl Trinitrate (GTN) and Nifedipine are widely used topical agents for anal fissure management. GTN acts as a nitric oxide donor, reducing sphincter tone via smooth muscle relaxation, though it is often associated with headaches. Nifedipine, a calcium channel blocker, lowers sphincter tone by inhibiting calcium influx into smooth muscle cells and has a more favorable side effect profile. Despite their widespread use, their comparative efficacy and safety remain a subject of debate.

This randomized controlled trial (RCT) aims to compare GTN and Nifedipine ointments in acute anal fissure treatment, evaluating symptom resolution, healing rates, and adverse effects to determine the optimal therapeutic choice.

Study Overview:

This double-blind, randomized, parallel-arm clinical trial will compare GTN and Nifedipine in patients with acute anal fissures. Participants will be allocated into:

GTN Group: Receiving either 0.2% or 0.4% GTN ointment, applied twice daily for four weeks.

Nifedipine Group: Receiving either 0.2% or 0.5% Nifedipine ointment, applied twice daily for four weeks.

The primary outcome is healing rate at four weeks, with secondary outcomes including pain reduction, side effects, patient satisfaction, and recurrence rates over six months.

Data Analysis:

Collected data will undergo statistical analysis using Chi-square tests, ANOVA, Kaplan-Meier survival analysis, and logistic regression modeling to identify treatment effectiveness and predictors of success.

Ethical Considerations:

The study is approved by the Federal Government Polyclinic Ethics Review Board, with written informed consent obtained from participants. All procedures comply with Good Clinical Practice (GCP) guidelines, and data confidentiality will be strictly maintained.

Expected Impact:

This study aims to refine treatment protocols for acute anal fissures, offering evidence-based guidance on the most effective and safest medical therapy, potentially reducing the need for surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria to be eligible for the study:
* Age 18 to 65 years (to exclude elderly patients with different treatment responses).
* Diagnosis of acute anal fissure based on clinical examination (symptom duration ≤6 weeks).
* Willingness to participate in the study and provide written informed consent.
* Availability for follow-up visits during the study period.
* No prior use of GTN or Nifedipine for anal fissure within the past one month.
* Presence of at least one of following symptoms: Anal pain, Bleeding during or after defecation and Difficulty in defecation

Exclusion Criteria:

* Participants will be excluded if they meet any of the following criteria:
* History of chronic anal fissure (>6 weeks duration) or prior anal fissure treatment within the past month.
* Pregnant or breastfeeding women.
* Known allergy or hypersensitivity to Glyceryl Trinitrate (GTN) or Nifedipine ointments.
* History of cardiovascular diseases or contraindications to GTN or Nifedipine (e.g., hypotension, severe heart disease).
* Presence of severe systemic diseases (e.g., uncontrolled diabetes, renal failure, autoimmune disorders) or conditions that may affect wound healing or medication tolerance.
* Use of other topical treatments for anal fissure within the past month.
* Secondary anal fissures associated with conditions e.g crohn's disease, tuberculosis, syphilis, HIV and other systemic diseases
* Previous anal surgery (including lateral internal sphincterotomy).
* History of recurrent anal fissures (>2 previous episodes in the past year).
* Inability to comply with study requirements or follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Healing Rate at 4 Weeks | 4 weeks
  The proportion of participants achieving complete epithelialization of the anal fissure on clinical examination at the end of four weeks.

SECONDARY OUTCOMES:
Change in Pain Scores (Visual Analog Scale [VAS]) | 4 weeks
  Reduction in pain scores from baseline to post-treatment, measured using the Visual Analog Scale (VAS), a 10-point scale ranging from 0 (no pain) to 10 (worst possible pain). Higher scores indicate greater pain severity.
Incidence and Severity of Adverse Effects | 4 weeks
  Assessment of drug-related side effects, including headache, dizziness, local irritation, and hypotension, recorded throughout the study duration.
Patient Satisfaction with Treatment ( Self-validated Patient Satisfaction Score) | 4 weeks
  Evaluation of patient-reported satisfaction with treatment outcomes, assessed using a structured questionnaire.
  Scoring System:
  Patient satisfaction is assessed using the Self-validated Patient Satisfaction Score, with responses recorded on a 5-point Likert scale. The scoring system is as follows:
  * Very satisfied = 5
  * Somewhat satisfied = 4
  * Neutral = 3
  * Somewhat dissatisfied = 2
  * Very dissatisfied = 1
    * Higher scores indicate greater patient satisfaction with treatment outcomes.
Time to Symptom Resolution | 4 weeks
  Duration until complete resolution of pain and cessation of rectal bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Ullah Khan, Consultant surgery, HOD, Study Chair — Federal Government Polyclinic (Postgraduate Medical Institute)
Locations (1):
- Federal Government Polyclinic (Postgraduate Medical Institute), Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, no final decision has been made regarding the sharing of individual participant data (IPD). Data sharing will be considered based on future research needs, ethical guidelines, and institutional policies. Any decision to share IPD will be made in compliance with data protection regulations and patient confidentiality standards.

REFERENCES:
- [Background] Mustafa NA, Cengiz S, Turkyilmaz S, Yucel Y. Comparison of topical glyceryl trinitrate ointment and oral nifedipine in the treatment of chronic anal fissure. Acta Chir Belg. 2006 Jan-Feb;106(1):55-8. doi: 10.1080/00015458.2006.11679834. PMID 16612915
- [Background] Wang C, Ni J, Xiong Y, Chen J, Li B, Xu L. The efficacy of diltiazem, glyceryl trinitrate, nifedipine, minoxidil, and lidocaine for the medical management of anal fissure: a systematic review and network meta-analysis of randomized controlled trials. Int J Surg. 2025 Apr 1;111(4):3020-3029. doi: 10.1097/JS9.0000000000002263. PMID 39878173
- [Background] Momayez Sanat Z, Mohammadi Ganjaroudi N, Mansouri M. The Effect of Topical Nifedipine versus Diltiazem on the Acute Anal Fissure: A Randomized Clinical Trial. Middle East J Dig Dis. 2023 Apr;15(2):121-125. doi: 10.34172/mejdd.2023.330. Epub 2023 Apr 30. PMID 37546514
- [Background] Shrestha SK, Thapa PB, Maharjan DK, Tamang TY. Effectiveness of 0.2% Glyceryl Trinitrate and 0.5% Nifedipine in the Treatment of Chronic Anal Fissure. JNMA J Nepal Med Assoc. 2017 Jan-Mar;56(205):149-152. PMID 28598453
- See also: Comparative Study of 0.2%GlycerylTrinitrate Ointment versus LateralInternal Sphincterotomy for Chronic Anal Fissure — https://www.researchgate.net/publication/377797898_Comparative_Study_of_Lateral_Internal_Sphincterotomy_versus_Local_04_Glyceryl_Trinitrate_Ointment_for_the_Treatment_of_Chronic_Anal_Fissure
- See also: FDA Approves GTN for Chronic Anal Fissure Pain — https://www.medscape.com/viewarticle/745118?form=fpf
- See also: Nifedipine 0.2% ointment is a topical calcium channel blocker used for anal fissure treatment, including in diabetic patients, by relaxing the anal sphincter and increasing blood flow. It is compounded with white petrolatum and has a USP beyond-use date — https://www.uspharmacist.com/article/nifedipine-02-ointment